CLINICAL TRIAL: NCT05832905
Title: Mobile and Wearable-assisted Case Management for Panic Disorder: An Observational Cohort Study Using Machine Learning and Explainable AI
Brief Title: Mobile-assisted Case Management for Panic Disorder
Acronym: MCM
Status: Completed | Type: Observational
Sponsor: En Chu Kong Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Principal Investigator, Chanhen Tsai, Attending Physician, En Chu Kong Hospital
Other Study IDs: EnChuKongH_MCM
Record Dates: First submitted 2023-03-26; First posted 2023-04-27 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Panic Disorder
Keywords: Wearables, Case Management, Mobile-assisted care
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experiment (observational) group with Mobile and Wearable-assisted Case Management (MCM): MCM involves the integration of mobile technology, such as smartphones and wearable devices, to supplement TAU. This approach is designed to provide additional support and monitoring to patients through the use of mobile applications and remote contact with healthcare professionals. In this study, MCM was implemented alongside TAU, with patients receiving pharmacotherapy, CBT, and mobile-assisted case management services. The MCM component consisted of regular contact with case managers via telephone and a dedicated mobile application.
  Interventions: Behavioral: Mobile and Wearable-assisted Case Management
- Control group (TAU): TAU refers to the standard care provided to patients with panic disorder, which typically includes a combination of pharmacotherapy and psychological or behavioral treatment. In the context of this study, TAU consisted of pharmacological interventions, such as prescribing anxiolytic or antidepressant medications, and psychological interventions, primarily Cognitive Behavioral Therapy (CBT). The administration of TAU was conducted by qualified healthcare professionals who followed established clinical guidelines and treatment protocols to ensure the appropriate management of panic disorder symptoms.
  Interventions: Behavioral: Mobile and Wearable-assisted Case Management

INTERVENTIONS:
Behavioral: Mobile and Wearable-assisted Case Management — The MCM group received case management and Mobile-and wearable recording. The actual intervention for Panic disorder, including pharmacotherapy or psychological treatment is the same as in MCM and TAU group

SUMMARY:
A panic attack (PA) is an intense form of anxiety accompanied by multiple somatic presentations, leading to frequent emergency department visits and impairing quality of life. A prediction model for PAs could help clinicians and patients monitor, control, and do early intervention for recurrent panic attacks, enabling more personalized treatment for panic disorder. This study aimed to provide a seven-day PA prediction model and determine the relationship between a future PA and various features, including physiological factors, anxiety and depressive factors, and air quality index. We will enroll 200 participants (150 participants join case management with wearables study, 50 participants join TAU group) with PD (DMS-5 and MINI interview). Participants used smartwatches (Garmin vivosmart 4) and mobile applications to collect their sleep, heart rate, activity level, anxiety, and depression scores (BDI, BAI, STAI-S, STAI-T, and PDSS-SR) in their real-life for a duration of one year. We also included air quality indexes from open data. To analyze these data, our team used six machine learning methods: random forests, decision trees, LDA, AdaBoost, XGBoost, and regularized greedy forests, or other deep learning methods.

DETAILED DESCRIPTION:
Participants enrollment Through primary psychiatrists' invitations, we will recruit 150 En Chu Kong Hospital psychiatric clinic PD participants and 50 patients from Mackay Memorial Hospital.

Inclusion criteria The inclusion criteria were 1) a primary diagnosis of PD by DSM-5, 2) more than 20 years old, and 3) an essential ability to navigate smartwatches and mobile phone applications. If participants did not fulfill criteria 3), we will invite them as the control group (i.e. TAU)

Exclusion criteria The exclusion criteria were 1) current substance abuse, 2) cardiopulmonary incapacity, 3) incapacity or limited mental capacity, and 4) acute suicidal ideation. This study required sufficient mental capacity on the part of participants to cooperate by wearing smartwatches continuously, properly maintaining the smartwatches, and completing regular, valid online questionnaires. Limited mental capacity implies that the participants have difficulties understanding, remembering, or using the information to make or communicate a decision. Our team evaluated participants' mental capacity during the diagnostic interview (DI), Mini International Neuropsychiatric Interview (MINI), and the informed consent process by certified psychiatrists and nurse practitioners. The information on acute suicidal ideation was from diagnostic interviews and questions from MINI part A and pre-assessment BDI.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of panic disorder by DSM5
2. More than 18 years old
3. An essential ability to navigate smartwatch and mobile phone applications

Exclusion Criteria:

1. Current substance abuse
2. Cardiopulmonary incapacity
3. Incapacity or limited mental capacity
4. Acute suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from outpatient clinics with a main diagnosis of Panic disorder
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
PDSS score | through study completion, an average of 1 year
  Panic severity score

SECONDARY OUTCOMES:
STAI score | through study completion, an average of 1 year
  The State-Trait Anxiety Inventory
BDI score | through study completion, an average of 1 year
  The Beck Depression Inventory II
BAI score | through study completion, an average of 1 year
  The Beck Anxiety Inventory

CONTACTS AND LOCATIONS:
Overall Officials: ECKIRB IRB, Principal Investigator — En Chu Kong Hostpial
Locations (1):
- En Chu Kong Hospital, Sanxia District, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsai CH, Chen PC, Liu DS, Kuo YY, Hsieh TT, Chiang DL, Lai F, Wu CT. Panic Attack Prediction Using Wearable Devices and Machine Learning: Development and Cohort Study. JMIR Med Inform. 2022 Feb 15;10(2):e33063. doi: 10.2196/33063. PMID 35166679